CLINICAL TRIAL: NCT04885270
Title: Phase III Clinical Trial of Intravenous Paclitaxel Plus Intraperitoneal Cisplatin for Neo-adjuvant Chemotherapy in Patients With Advanced Ovarian Cancer
Brief Title: Paclitaxel i.v. Plus Cisplatin i.p for NACT in Patients With Advanced Ovarian Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Rutie Yin, Professor, West China Second University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WestChinaSUH2020076
Record Dates: First submitted 2021-04-27; First posted 2021-05-13 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Epithelial Carcinoma, Ovarian; Neoadjuvant Chemotherapy
Keywords: intraperitoneal chemotherapy; neoadjuvant chemotherapy; Epithelial ovarian cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm i.p (Experimental): paclitaxel i.v. and cisplatin i.p.
  Interventions: Drug: cisplatin i.p.

INTERVENTIONS:
Drug: cisplatin i.p. — paclitaxel 135 mg/m2 i.v. and cisplatin 75 mg/m2 i.p. on day 1
  Other Names: intraperitoneal cisplatin

SUMMARY:
To test the effect of intravenous paclitaxel plus intraperitoneal cisplatin for neo-adjuvant chemotherapy in patients with advanced ovarian cancer, the investigators conducted a phase III single arm clinical trial. Included patients will receive interval debulking surgery after 2-6 cycles neoadjuvant chemotherapy based on the clinical judgment of the gynecologic oncologist. Six cycles of chemotherapy will conducted after surgery. And the neoadjuvant chemotherapy is as follows: paclitaxel 135 mg/m2 i.v. and cisplatin 75 mg/m2 i.p. on day 1. The primary end point is optimal debulking rates. the investigators also will evaluate effect on parameters of volume of ascites, tumor size, duration of surgery, hemorrhage, hospitalizations and postoperative complication etc. After comparing with data published online, the investigators will try to find out if paclitaxel i.v. plus cisplatin i.p. is a superior neoadjuvant chemotherapy for advanced ovarian carcinoma.

DETAILED DESCRIPTION:
1. BACKGROUND AND INTRODUCTION Epithelial ovarian cancer (EOC) is the leading cause of death from gynecologic malignancy in the developed world with the majority of women presenting with stage III/IV disease. Most patients with advanced-stage cancer will eventually experience recurrence and die as a result of the disease. Therefore, more effective therapies are needed in the treatment of this aggressive cancer.

   After the results of the Gynecologic Oncology Group trial (GOG-152) (NCT00002568) the investigatorsre published, interval debulking surgery was no longer recommended for patients in whom optimal cytoreduction was not achieved despite a maximal effort at primary debulking surgery[1]. The use of neoadjuvant chemotherapy (NACT) before a definitive debulking attempt is increasingly used in advanced EOC based on two RCTs (EORTC55971 and CHORUS) which demonstrated non-inferiority and lothe investigatorsr perioperative morbidity compared with primary surgery follothe investigatorsd by chemotherapy[2, 3]. But what is the preferred chemotherapy regimen for women who will receive NACT is still a question[4].

   Evidence from the peritoneal dialysis literature suggests that the peritoneal permeability of a number of hydrophilic anticancer drugs may be considerably less than plasma clearance. Pharmacokinetic calculations indicate that such drugs administered i.p.(intraperitoneal chemotherapy,i.p.) in large volumes are expected to maintain a significantly greater concentration in the peritoneal space than in the plasma. Prior studies have reported on the pharmacologic advantage of delivering cisplatin i.p., with a 20-fold higher concentration in the i.p. space compared with that measured in plasma after i.v. administration[5]. This concentration difference offers a potentially exploitable biochemical advantage in the treatment of patients with presumed microscopic residual ovarian cancer confined to the peritoneal cavity[6]. In addition, i.p. therapy allows for continuous and prolonged exposure of high drug concentrations with lothe investigatorsr peak plasma levels over time[7].

   Three randomized clinical trials (RCTs) and a meta-analysis had demonstrated improved survival for women with stage III EOC who received a combination of i.v. and i.p. chemotherapy following optimal, primary debulking surgery[8-10]. GOG 172 confirmed a continued benefit for women who had received the experimental arm[11]. OV21/PETROC proved in women with stage IIIC or IVA EOC treated with NACT and optimal debulking surgery, i.p. carboplatin-based chemotherapy is the investigatorsll tolerated and associated with an improved PD9 (9-month progressive disease rate) compared with i.v. carboplatin-based chemotherapy. But there is no RCT focused on the role of i.p. in NACT[12].

   From the retrospective data in our institution (not published yet), compared with intravenous paclitaxel plus carboplatin, intravenous paclitaxel plus i.p. cisplatin shothe investigatorsd more effective in NACT, and side effects like nausea and vomiting are acceptable and manageable, moreover, with lothe investigatorsr bone marrow suppression rate. To determine the role of i.p. cisplatin in NACT the investigators desiged a RCT to compare optimal debulking rates and progression-free survival (PFS) in women with stage IIIc or IV epithelial ovarian carcinoma after treated with NACT using intravenous paclitaxel plus carboplatin and intravenous paclitaxel plus i.p. cisplatin.
2. OBJECTIVES OF THE TRIAL To test effect of intravenous paclitaxel plus intraperitoneal cisplatin for neo-adjuvant chemotherapy in patients with advanced ovarian cancer
3. TRIAL DESIGN. Treatment: paclitaxel 135 mg/m2 i.v. and cisplatin 75 mg/m2 i.p. on day 1

   Principal surgeon:

   Only senior surgeons will be allothe investigatorsd to have the responsibility for the surgery. Each senior surgeon will follow carefully the guideline for surgery.

   Cycle of chemotherapy:

   Surgery may be performed after 2-6 cycles based on the clinical judgment of the gynecologic oncologist. Six cycles of chemotherapy will conducted after surgery.
4. THERAPEUTIC REGIMENS Interval debulking surgery should be performed within 6 the investigatorseks after course 2-6 in all patients with response or stable disease. If this time limit is not met the patient has to be excluded from this protocol. Follothe investigatorsd by 6 courses of chemotherapy within 3 the investigatorseks after surgery.

   Regimens: paclitaxel 135 mg/m2 i.v. and cisplatin 75 mg/m2 i.p. on day 1
5. ENDPOINT OF THIS STUDY First stage

Primary end point:

Optimal debulking rates

* Optimal cytoreduction was defined as largest residual tumor nodule not greater than 1 cm in maximal diameter at the completion of the primary operation.

Secondary end points:

Volume of ascites Tumor size Duration of surgery, hemorrhage, hospitalizations Postoperative complication (infection, venous complications, hospitalization etc.) AEs of chemotherapy

*Upper abdomen surgical procedures the investigatorsre defined as splenectomy, pancreatectomy, gallbladder resection, liver resection, diaphragmatic resection.

Second stage Primary end point Progression free survival (PFS) Secondary end points Overall survival (OS)

ELIGIBILITY:
Inclusion Criteria:

1. Preferentially biopsy proven Stage IIIc or IV epithelial ovarian carcinoma, or peritoneal or fallopian tube carcinoma (the presence of metastases outside the pelvis measuring at least 2 cm in diameter (as noted during diagnostic laparoscopy or laparotomy or on computed tomography [CT]),with a low likelihood of achieving cytoreduction to, 1 cm (ideally to no visible disease). Or women who have a high perioperative risk profile.
2. Fine needle aspiration (FNA) showing an adenocarcinoma and cytopathology from ascites or pleural effusion is acceptable under the following conditions:

   the patient has a pelvic (ovarian) mass, AND omental cake or other metastasis larger than 2 cm in the upper abdomen and/or regional lymphnode metastasis irrespective of size or stage IV AND serum CA125/CEA ratio > 25. If the serum CA125/CEA ratio is < 25, a barium enema (or colonoscopy) and gastroscopy (or radiological examination of the stomach) should be negative for the presence of a primary tumor (< 6 weeks before randomization), and normal mammography (< 6 weeks).
3. WHO performance status of 0, 1, or 2.
4. No other serious disabling diseases contraindicating for cytoreductive surgery or platin based chemotherapy.
5. No other prior primary malignancies, except for carcinoma in situ of the cervix and basal carcinoma of the skin.
6. No clinical evidence of brain or leptomeningeal metastases.
7. Adequate hematological, renal and hepatic function to permit platin-paclitaxel based chemotherapy: WBC > 3.0 x 109/L, N >1.5 x 109/L, platelets > 100 x 109/L, serum creatinine < 1.25 x upper normal range, serum bilirubin < 1.25 x upper normal range.
8. Absence of any psychological, familial, sociological or geographical condition potentially preventing compliance with the study protocol and follow-up schedule; those conditions should be assessed with the patient before registration in the trial.
9. Before patient registration/randomization, informed consent must be obtained and documented according to national and local regulatory requirements and the local rules followed in the institution.

Exclusion Criteria:

1. serious disabling diseases that would contraindicate primary cytoreductive surgery or platinumbased chemotherapy
2. mucinous or borderline histology, extensive intra-abdominal adhesions, bowel obstruction or unresolved>grade 2 peripheral neuropathy.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-08-04 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Optimal debulking rates | up to 18 weeks
  Optimal cytoreduction was defined as largest residual tumor nodule not greater than 1 cm in maximal diameter at the completion of the primary operation.
PFS | Progression free survival (PFS) will be measured from the date enrollment to the first documented date of progression, or death, whichever occurs first, assessed up to 36 months.
  Progression free survival

SECONDARY OUTCOMES:
OS | Overall survival (OS) will be measured from the date of enrollment to the date of death, whatever the cause, assessed up to 36 months.
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- West China Second University Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rose PG, Nerenstone S, Brady MF, Clarke-Pearson D, Olt G, Rubin SC, Moore DH, Small JM; Gynecologic Oncology Group. Secondary surgical cytoreduction for advanced ovarian carcinoma. N Engl J Med. 2004 Dec 9;351(24):2489-97. doi: 10.1056/NEJMoa041125. PMID 15590951
- [Background] Kehoe S, Hook J, Nankivell M, Jayson GC, Kitchener H, Lopes T, Luesley D, Perren T, Bannoo S, Mascarenhas M, Dobbs S, Essapen S, Twigg J, Herod J, McCluggage G, Parmar M, Swart AM. Primary chemotherapy versus primary surgery for newly diagnosed advanced ovarian cancer (CHORUS): an open-label, randomised, controlled, non-inferiority trial. Lancet. 2015 Jul 18;386(9990):249-57. doi: 10.1016/S0140-6736(14)62223-6. Epub 2015 May 19. PMID 26002111
- [Background] Vergote I, Trope CG, Amant F, Kristensen GB, Ehlen T, Johnson N, Verheijen RH, van der Burg ME, Lacave AJ, Panici PB, Kenter GG, Casado A, Mendiola C, Coens C, Verleye L, Stuart GC, Pecorelli S, Reed NS; European Organization for Research and Treatment of Cancer-Gynaecological Cancer Group; NCIC Clinical Trials Group. Neoadjuvant chemotherapy or primary surgery in stage IIIC or IV ovarian cancer. N Engl J Med. 2010 Sep 2;363(10):943-53. doi: 10.1056/NEJMoa0908806. PMID 20818904
- [Background] Wright AA, Bohlke K, Armstrong DK, Bookman MA, Cliby WA, Coleman RL, Dizon DS, Kash JJ, Meyer LA, Moore KN, Olawaiye AB, Oldham J, Salani R, Sparacio D, Tew WP, Vergote I, Edelson MI. Neoadjuvant Chemotherapy for Newly Diagnosed, Advanced Ovarian Cancer: Society of Gynecologic Oncology and American Society of Clinical Oncology Clinical Practice Guideline. J Clin Oncol. 2016 Oct 1;34(28):3460-73. doi: 10.1200/JCO.2016.68.6907. Epub 2016 Aug 8. PMID 27502591
- [Background] Lopez JA, Krikorian JG, Reich SD, Smyth RD, Lee FH, Issell BF. Clinical pharmacology of intraperitoneal cisplatin. Gynecol Oncol. 1985 Jan;20(1):1-9. doi: 10.1016/0090-8258(85)90118-0. PMID 4038390
- [Background] Dedrick RL, Myers CE, Bungay PM, DeVita VT Jr. Pharmacokinetic rationale for peritoneal drug administration in the treatment of ovarian cancer. Cancer Treat Rep. 1978 Jan;62(1):1-11. PMID 626987
- [Background] Tummala MK, Alagarsamy S, McGuire WP. Intraperitoneal chemotherapy: standard of care for patients with minimal residual stage III ovarian cancer? Expert Rev Anticancer Ther. 2008 Jul;8(7):1135-47. doi: 10.1586/14737140.8.7.1135. PMID 18588458
- [Background] Alberts DS, Liu PY, Hannigan EV, O'Toole R, Williams SD, Young JA, Franklin EW, Clarke-Pearson DL, Malviya VK, DuBeshter B. Intraperitoneal cisplatin plus intravenous cyclophosphamide versus intravenous cisplatin plus intravenous cyclophosphamide for stage III ovarian cancer. N Engl J Med. 1996 Dec 26;335(26):1950-5. doi: 10.1056/NEJM199612263352603. PMID 8960474
- [Background] Armstrong DK, Bundy B, Wenzel L, Huang HQ, Baergen R, Lele S, Copeland LJ, Walker JL, Burger RA; Gynecologic Oncology Group. Intraperitoneal cisplatin and paclitaxel in ovarian cancer. N Engl J Med. 2006 Jan 5;354(1):34-43. doi: 10.1056/NEJMoa052985. PMID 16394300
- [Background] Markman M, Bundy BN, Alberts DS, Fowler JM, Clark-Pearson DL, Carson LF, Wadler S, Sickel J. Phase III trial of standard-dose intravenous cisplatin plus paclitaxel versus moderately high-dose carboplatin followed by intravenous paclitaxel and intraperitoneal cisplatin in small-volume stage III ovarian carcinoma: an intergroup study of the Gynecologic Oncology Group, Southwestern Oncology Group, and Eastern Cooperative Oncology Group. J Clin Oncol. 2001 Feb 15;19(4):1001-7. doi: 10.1200/JCO.2001.19.4.1001. PMID 11181662
- [Background] Tewari D, Java JJ, Salani R, Armstrong DK, Markman M, Herzog T, Monk BJ, Chan JK. Long-term survival advantage and prognostic factors associated with intraperitoneal chemotherapy treatment in advanced ovarian cancer: a gynecologic oncology group study. J Clin Oncol. 2015 May 1;33(13):1460-6. doi: 10.1200/JCO.2014.55.9898. Epub 2015 Mar 23. PMID 25800756
- [Background] Provencher DM, Gallagher CJ, Parulekar WR, Ledermann JA, Armstrong DK, Brundage M, Gourley C, Romero I, Gonzalez-Martin A, Feeney M, Bessette P, Hall M, Weberpals JI, Hall G, Lau SK, Gauthier P, Fung-Kee-Fung M, Eisenhauer EA, Winch C, Tu D, MacKay HJ. OV21/PETROC: a randomized Gynecologic Cancer Intergroup phase II study of intraperitoneal versus intravenous chemotherapy following neoadjuvant chemotherapy and optimal debulking surgery in epithelial ovarian cancer. Ann Oncol. 2018 Feb 1;29(2):431-438. doi: 10.1093/annonc/mdx754. PMID 29186319